CLINICAL TRIAL: NCT00850993
Title: A Phase 2b, Multicenter, Single-dose, Blinded, Randomized, Placebo-controlled, Dose-escalation, Safety and Efficacy Trial of Stannsoporfin in Neonates With Hyperbilirubinemia
Brief Title: A Safety and Efficacy Trial of Stannsoporfin in Neonates With Hyperbilirubinemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: To redefine study population
Sponsor: InfaCare Pharmaceuticals Corporation, a Mallinckrodt Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 64,185-202; 2009-017434-45 (EudraCT Number)
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2014-08

CONDITIONS: Hyperbilirubinemia, Neonatal
Keywords: Hemolysis
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hemolysis | interventions — tin mesoporphyrin; Sodium Chloride; Phototherapy

STUDY DESIGN:
Intervention Model Description: Sequential experimental cohorts are run in parallel with placebo controls.
Who Masked: Participant, Investigator
Masking Description: Clinical personnel at the site (including investigator, study coordinator and central cardiologist) were blinded to treatment group.
  The research pharmacy and the health care provider responsible for giving the injection to patients knew what the treatment was (they were not blinded).
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1: Stannsoporfin 1.5 mg/kg (Experimental): Participants receive a single dose of 1.5 mg/kg by intramuscular (IM) injection, along with PhotoTherapy (PT) if and when needed.
  Interventions: Drug: Stannsoporfin; Other: PhotoTherapy (as needed)
- Cohort 2: Stannsoporfin 3.0 mg/kg (Experimental): Participants receive a single dose of 3.0 mg/kg by intramuscular (IM) injection, along with PT if and when needed.
  Interventions: Drug: Stannsoporfin; Other: PhotoTherapy (as needed)
- Cohort 3: Stannsoporfin 4.5 mg/kg (Experimental): Participants receive a single dose of 4.5 mg/kg by intramuscular (IM) injection, along with PT if and when needed.
  Interventions: Drug: Stannsoporfin; Other: PhotoTherapy (as needed)
- Cohort 4: Placebo (Placebo Comparator): Participants receive a single dose of placebo (sterile saline solution) by IM injection, along with PT if and when needed.
  Interventions: Other: Placebo; Other: PhotoTherapy (as needed)

INTERVENTIONS:
Drug: Stannsoporfin — Stannsoporfin administered as a single IM injection
  Other Names: Experimental product
  Arms: Cohort 1: Stannsoporfin 1.5 mg/kg; Cohort 2: Stannsoporfin 3.0 mg/kg; Cohort 3: Stannsoporfin 4.5 mg/kg
Other: Placebo — Placebo (sterile saline solution) administered as a single IM injection
  Other Names: Saline
  Arms: Cohort 4: Placebo
Other: PhotoTherapy (as needed) — PT standard care administered as needed, based on bilirubin levels throughout the treatment period
  Other Names: PT

SUMMARY:
It is a normal process in the human body for red blood cells to die, which makes bilirubin.

Bilirubin is cleared away through the liver.

Some babies are born with livers that don't work well enough yet, or their red blood cells are dying too fast, so the baby looks yellow (jaundice).

This means there is too much bilirubin in the body. It can be dangerous if a baby's bilirubin gets too high.

Phototherapy is what they call the lights they shine on newborn babies to help the liver get rid of bilirubin.

This study tests an experimental drug to see if it can reduce how much bilirubin is being made in the first place.

DETAILED DESCRIPTION:
The purpose of this study is to determine if an experimental drug, stannsoporfin, is safe and effective in the treatment of hyperbilirubinemia in hemolyzing neonates.

ELIGIBILITY:
Inclusion Criteria:

Babies may only participate if they meet all the following criteria:

* Is a term or late preterm baby
* Is at risk for protocol-defined hemolytic disease
* Weighs at least 2500 g (5.5 lbs)
* Has total serum bilirubin (TSB) a specified amount lower than the phototherapy threshold for the age
* Has parents/guardians who are willing to follow light precautions and sign informed consent

Exclusion Criteria:

The following criteria will make a baby not eligible to participate:

* Needs medications that may prolong the QT interval
* Has family history or risk factors for Long QT Syndrome, Sudden Infant Death Syndrome, or Porphyrias
* Has an Apgar score of 6 or below at age 5 minutes
* Has abnormalities or infections (in mother or child) that per protocol or in the opinion of the investigator may compromise the safety and well-being of the baby or analysis of study results

Ages: 1 Minute to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt
Locations (23):
- United States (9):
  - Arrowhead Regional Med Center, Colton, California
  - UCSD Medical Center, San Diego, California
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii
  - University of Louisville, Louisville, Kentucky
  - Westchester Medical Center, Valhalla, New York
  - ECU Brody School of Medicine, Greenville, North Carolina
  - St. Vincent Mercy Children's Hospital, Toledo, Ohio
  - Drexel University College of Medicine, Clinical Research Group, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
- Poland (3):
  - Jan Bizel University Hospital No. 2; Department of Neonatal, Preemies and Neonatal Intensive Care, Bydgoszcz
  - Research Institute of Polish Mother's Health Center, Lodz
  - Neonatal Department Warsaw Medical University, Warsaw
- Spain (6):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Vall D´Hebrón, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Doce de Octubre, Madrid
  - Hospital La Paz, Madrid
  - University Hospital Santiago de Compostela-L Coruna, Santiago de Compostela
- Ukraine (5):
  - Municipal Medical Institution "Regional pediatric clinical hospital #1", Department of pathology of the newborns; Bukovynian State Medical University, Department of Pediatrics and Children's Infectious Diseases, Chernivtsi
  - National Pediatric Specialized Hospital "OHMATDYT"., Kiev
  - State Institution "Institute of Pediatrics, Obstetrics and Gynecology of the Academy of Medical Science of the Ukraine", Neonatology Department, Kiev
  - Municipal Institution "Odessa regional clinical hospital", Department of pathology of the newborns and premature infants; Odessa State Medical University; Chair of Pediatrics #1 and Neonatology, Odesa
  - Vinnytsia regional pediatric hospital, Department of pathology of the newborns, Vinnytsia National Medical University named after M.I.Pirogov, Chair of Pediatrics #1, Vinnitsa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-eight (58) babies were enrolled before the trial was prematurely terminated due to cancellation.
Pre-assignment Details: Because the cohorts were run sequentially, and the trial was cancelled before they were all enrolled, Cohort 3 enrolled only 8 compared to 15 in Cohort 4.
Groups:
- Cohort 1: Stannsoporfin 1.5 mg/kg: 1.5 mg/kg stannsoporfin (with phototherapy as needed)
- Cohort 2: Stannsoporfin 3.0 mg/kg: 3.0 mg/kg stannsoporfin (with phototherapy as needed)
- Cohort 3: Stannsoporfin 4.5 mg/kg: 4.5 mg/kg stannsoporfin (with phototherapy as needed)
- Cohort 4: Placebo Control: Placebo control was sterile saline solution (with phototherapy as needed)
Period: Overall Study
Arm/Group | Cohort 1: Stannsoporfin 1.5 mg/kg | Cohort 2: Stannsoporfin 3.0 mg/kg | Cohort 3: Stannsoporfin 4.5 mg/kg | Cohort 4: Placebo Control
Started | 17 | 18 | 8 | 15
Safety | 17 | 18 | 8 | 15
Intent-to-treat | 17 | 18 | 8 | 15
Received Phototherapy | 3 | 6 | 2 | 8
Per Protocol | 10 | 13 | 5 | 13
Completed | 16 | 18 | 8 | 14
Not Completed | 1 | 0 | 0 | 1
Not completed — Parent/Guardian Voluntarily Withdrew | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Stannsoporfin 1.5 mg/kg | Cohort 2: Stannsoporfin 3.0 mg/kg | Cohort 3: Stannsoporfin 4.5 mg/kg | Cohort 4: Placebo Control | Total
Number analyzed (Participants) | 17 | 18 | 8 | 15 | 58
Age, Customized [Count of Participants; unit: Participants] — Gestational Age, Categorical
  Participants
    35 through 37 Weeks | 2 | 0 | 1 | 3 | 6
    38 Weeks and Above | 15 | 18 | 7 | 12 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 6 | 7 | 29
  Male | 7 | 12 | 2 | 8 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 6 | 4 | 21
  Not Hispanic or Latino | 12 | 12 | 2 | 11 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 4 | 3 | 0 | 4 | 11
  Black or African American | 5 | 2 | 0 | 2 | 9
  White | 7 | 7 | 6 | 3 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 2 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Adjusted Total Serum Bilirubin (TSB) From Baseline to 48 Hours After Treatment.
Description: The adjusted TSB is a calculation of the percentage difference of the TSB level from the age-specific threshold for PT initiation per the American Academy of Pediatrics (AAP) Guidelines, ie, an indication of the distance below the PT threshold at the time [(TSB - PT threshold/PT threshold) x 100%).
Time Frame: Baseline, 48 hours
Population: Intent-to-treat population (ITT)
Measure: Median (Full Range); unit: percentage difference from PT threshold
Groups:
- Placebo Control: Sterile saline solution (with phototherapy as needed)
Arm/Group | Cohort 1: Stannsoporfin 1.5 mg/kg | Cohort 2: Stannsoporfin 3.0 mg/kg | Cohort 3: Stannsoporfin 4.5 mg/kg | Placebo Control
Number analyzed (Participants) | 17 | 18 | 8 | 15
percentage difference from PT threshold | -12.30 [-55.7 to 0.3] | -9.05 [-54.8 to 12.0] | -19.95 [-59.0 to -5.0] | -5.7 [-42.1 to 22.2]
Statistical Analysis 1: Comparison: Cohort 1: Stannsoporfin 1.5 mg/kg vs Placebo Control; Last Observation Carry Forward (LOCF) is used to impute missing post-baseline TSB. Least-squares means are from an ANCOVA model for adjusted TSB with treatment and gestational age as fixed effects and baseline adjusted TSB as a covariate. TSB is calculated as [(TSB - Phototherapy(PT) threshold)/ PT threshold ] X 100%; Test type: Other — Pairwise comparison for each Stannsoporfin treatment group versus placebo; p = 0.040, ANCOVA; LS Mean Difference = -13.45, 95% CI 2-sided [-26.27 to -0.62]
Statistical Analysis 2: Comparison: Cohort 2: Stannsoporfin 3.0 mg/kg vs Placebo Control; Test type: Other; p = 0.117, ANCOVA; LS Mean Difference = -10.02, 95% CI 2-sided [-22.61 to 2.58]
Statistical Analysis 3: Comparison: Cohort 3: Stannsoporfin 4.5 mg/kg vs Placebo Control; Test type: Other; p = 0.057, ANCOVA; LS Mean Difference = -14.93, 95% CI 2-sided [-30.31 to 0.44]

2. Primary Outcome: Change From Baseline in Total Serum Bilirubin (TSB) at 48 Hours (ITT Population
Description: Total bilirubin in blood serum was measured at baseline and at 48 hours after the shot. Change from baseline is calculated by subtracting the amount at baseline from the amount at 48 hours. Lower numbers are better.
Time Frame: Baseline, 48 hrs
Population: Intention-to-treat
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Cohort 1: Stannsoporfin 1.5 mg/kg | Cohort 2: Stannsoporfin 3.0 mg/kg | Cohort 3: Stannsoporfin 4.5 mg/kg | Placebo Control
Number analyzed (Participants) | 17 | 18 | 8 | 15
mg/dL
  at Baseline | 7.80 [4.3 to 12.0] | 8.45 [5.5 to 10.4] | 9.35 [6.4 to 12.8] | 8.00 [4.6 to 11.9]
  at 48 hours | 10.90 [3.3 to 13.5] | 11.65 [4.2 to 14.1] | 10.35 [5.6 to 13.4] | 11.90 [8.1 to 15.8]
  Change from Baseline at 48 hours | 2.70 [-4.5 to 5.2] | 2.94 [-3.4 to 6.2] | 1.45 [-3.4 to 3.6] | 3.70 [-0.2 to 8.7]
Statistical Analysis 1: Comparison: Cohort 1: Stannsoporfin 1.5 mg/kg vs Placebo Control; Last Observation Carry Forward (LOCF) is used to impute missing post-baseline TSB. Analysis of covariance (ANCOVA) is conducted for TSB including treatment and gestational age as fixed effects and baseline TSB as a covariate. Least-squares means (LS means) and standard errors (SEM) are estimated for each treatment group and placebo. LS mean difference, 95% Confidence Interval, and p-value are estimated based on LS mean difference between each stannsoporfin group and placebo; Test type: Other — Pairwise comparison for Change from Baseline at 48 hours (Row 3) for Stannsoporfin treatment group versus placebo; p = 0.061, ANCOVA; LS Mean Difference = -1.81, 95% CI 2-sided [-3.71 to 0.09]
Statistical Analysis 2: Comparison: Cohort 2: Stannsoporfin 3.0 mg/kg vs Placebo Control; [analysis description as in outcome 2, analysis 1]; Test type: Other — Pairwise comparison for Change from Baseline at 48 hours (Row 3) for Stannsoporfin treatment group versus placebo; p = 0.163, ANCOVA; LS Mean Difference = -1.34, 95% CI 2-sided [-3.24 to 0.56]
Statistical Analysis 3: Comparison: Cohort 3: Stannsoporfin 4.5 mg/kg vs Placebo Control; [analysis description as in outcome 2, analysis 1]; Test type: Other — Pairwise comparison for Change from Baseline at 48 hours (Row 3) for Stannsoporfin treatment group versus placebo; p = 0.028, ANCOVA; LS Mean Difference = -2.63, 95% CI 2-sided [-4.97 to -0.3]

ADVERSE EVENTS:
Time Frame: 30 days
Description: All adverse events were collected by the investigator except jaundice and hyperbilirubinemia after the first amendment.
Arm/Group | Cohort 1: Stannsoporfin 1.5 mg/kg | Cohort 2: Stannsoporfin 3.0 mg/kg | Cohort 3: Stannsoporfin 4.5 mg/kg | Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18 | 0/8 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/18 | 1/8 | 2/15
Other Adverse Events (participants affected / at risk) | 8/17 | 10/18 | 3/8 | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Stannsoporfin 1.5 mg/kg (N=17) | Cohort 2: Stannsoporfin 3.0 mg/kg (N=18) | Cohort 3: Stannsoporfin 4.5 mg/kg (N=8) | Placebo Control (N=15)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Stannsoporfin 1.5 mg/kg (N=17) | Cohort 2: Stannsoporfin 3.0 mg/kg (N=18) | Cohort 3: Stannsoporfin 4.5 mg/kg (N=8) | Placebo Control (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Jaundice (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood sodium increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carbon dioxide decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne infantile (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash neonatal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
It should be noted that the study was discontinued before enrollment of the full 4.5 mg/kg cohort,and therefore, the stannsoporfin 4.5 mg/kg treatment group included 8 patients and the placebo group included 15 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days